CLINICAL TRIAL: NCT02508844
Title: The POP-study: Effect of Probiotics on Weight, Microbiota and Glucose Tolerance in Obese Pregnant Women and Their Newborn - a Randomized, Double-blind Placebo Controlled Trial With Vivomixx®
Brief Title: Effect of Probiotics (Vivomixx®) on Weight, Microbiota and Glucose Tolerance in Obese Pregnant Women and Their Newborn
Acronym: POP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, MD, clinical associate professor, Ph.D., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2-2014-076
Record Dates: First submitted 2015-05-11; First posted 2015-07-27 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy; Obesity; Gestational Diabetes Mellitus
Keywords: Probiotics; Vivomixx®; Microbiota
MeSH Terms: conditions — Obesity; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vivomixx® (Experimental): Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, Lactobacillus bulgaricus and Streptococcus thermophilus
  Interventions: Dietary Supplement: Vivomixx®
- Placebo (Placebo Comparator): microcrytalline cellulose, magnesium stearate and silicon dioxide.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — probiotics intake (four capsules of Vivomixx®; total of 450 billion CFU/day) from gestational age 14-20 until delivery
  Arms: Vivomixx®
Dietary Supplement: Placebo — Four capsules/day from gestational age 14-20 until delivery. The placebo capsule contains microcrytalline cellulose, magnesium stearate and silicon dioxide.
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate if the probiotics Vivomixx® can affect gestational weight gain, microbiota and pregnancy complications in pregnant obese women and birth weight body composition of their infants.

DETAILED DESCRIPTION:
Accumulating evidence indicates that the gut microbiota plays a significant role in obesity and because the "ideal" composition of the gut microbiota remains poorly understood, modulation of the gut microbiota composition represents a potentially attractive treatment option against excessive gestational weight gain and adverse outcomes for obese pregnant women and their newborn. Dietary supplements in the form of probiotics could be an efficient treatment for controlling weight gain in pregnancy by inducing changes in the gut microbiota and could have influence on infant's microbiota, which could have important implications for infant development and health.

A pilot study including 50 obese pregnant nulliparous with BMI between 30-35 kg/m2 will, after accepting participation, be randomized to receive daily placebo or probiotics (four capsules of Vivomixx®; total of 450 billion CFU/day) from gestational age 14-20 until delivery. The infants will be followed until 9 months of age. Shortly after birth, tissue composition will be measured in the infants by DEXA-scanning. The women will be monitored by weight, blood-, fecal- and urine samples, diet questionnaires and hospital record review. Vivomixx® is a probiotic mixture of 8 probiotic strains, (Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, Lactobacillus bulgaricus and Streptococcus thermophilus).

This is the first pilot study in which the probiotic Vivomixx® are added in a randomized fashion to the standard of care in obese pregnant women. 50 pregnant women are planned to be included. The aim of this group size is to clarify the feasibility, compliance and to estimate parameters such as the standard deviation which will be used in a sample size calculation for a full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 and ≤35 kg/m2- calculated from pre-pregnancy weight
* Primiparous singleton pregnancy
* Able to read and speak Danish
* Normal ultrasound scan of the fetus at gestational age 12-14
* Oral glucose tolerance test at gestational age 14-20

Exclusion Criteria:

* Pregnancy at > 20 weeks gestation at recruitment
* Pre-gestational diabetes or other serious diseases
* Multiple pregnancy
* Previous bariatric surgery
* Ingestion of probiotics < 1 month before the inclusion or ingestion of other kinds of probiotics than the study probiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | week 36-37 of pregnancy
  weight at gestational age 36-37-weeks minus self-reported pre-pregnancy weight
Change in glucose levels (Oral glucose tolerance test) | baseline (week 14-20) and 27-30 of pregnancy

SECONDARY OUTCOMES:
Change in fecal microbiota | baseline (week 14-20) and week 36-37 of pregnancy
Amount of fat tissue in the newborn infant | at birth
  examined by a DEXA-scanning
Change in HbA1c | baseline (week 14-20) and week 36-37 of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD, PhD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Halkjaer SI, de Knegt VE, Kallemose T, Jensen JB, Cortes D, Gluud LL, Wewer Albrechtsen NJ, Petersen AM. No effect of multi-strain probiotic supplementation on metabolic and inflammatory markers and newborn body composition in pregnant women with obesity: Results from a randomized, double-blind placebo-controlled study. Nutr Metab Cardiovasc Dis. 2023 Dec;33(12):2444-2454. doi: 10.1016/j.numecd.2023.07.030. Epub 2023 Jul 28. PMID 37580231
- [Derived] Halkjaer SI, de Knegt VE, Lo B, Nilas L, Cortes D, Pedersen AE, Mirsepasi-Lauridsen HC, Andersen LO, Nielsen HV, Stensvold CR, Johannesen TB, Kallemose T, Krogfelt KA, Petersen AM. Multistrain Probiotic Increases the Gut Microbiota Diversity in Obese Pregnant Women: Results from a Randomized, Double-Blind Placebo-Controlled Study. Curr Dev Nutr. 2020 May 27;4(7):nzaa095. doi: 10.1093/cdn/nzaa095. eCollection 2020 Jul. PMID 32617453
- [Derived] Halkjaer SI, Nilas L, Carlsen EM, Cortes D, Halldorsson TI, Olsen SF, Pedersen AE, Krogfelt KA, Petersen AM. Effects of probiotics (Vivomixx(R)) in obese pregnant women and their newborn: study protocol for a randomized controlled trial. Trials. 2016 Oct 11;17(1):491. doi: 10.1186/s13063-016-1617-5. PMID 27724923